CLINICAL TRIAL: NCT03929588
Title: A Clinical Validation Study to Evaluate the Performance of a Hand-held Device Supported by a Mobile Application Compared With Standard Eye Care Diagnostic Devices in Measuring Refractive Error of the Eye
Brief Title: Study of a Hand-held Device Plus Mobile App Versus Standard Eye Care Devices in Measuring Refractive Error of the Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EyeQue Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: EYEQUE - 001
Record Dates: First submitted 2019-04-22; First posted 2019-04-29 (Actual); Results first posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-02

CONDITIONS: Refractive Errors; Astigmatism
Keywords: myopia; hyperopia
MeSH Terms: conditions — Refractive Errors; Astigmatism; Myopia; Hyperopia

STUDY DESIGN:
Intervention Model Description: All enrolled subjects will have measurements with the phoropter, autorefractor and handheld device plus mobile app.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Refraction with a Hand-held Device Supported by Mobile App. (Experimental): BCVA with handheld device with app.
  Interventions: Device: Phoropter; Device: Autorefractor
- Manual Refraction (Active Comparator): BCVA with phoropter
  Interventions: Device: Hand-held device supported by a mobile application
- Automated Refraction (Active Comparator): BCVA with autorefractoer
  Interventions: Device: Hand-held device supported by a mobile application

INTERVENTIONS:
Device: Hand-held device supported by a mobile application — Hand-held device supported by a mobile application to obtain refractive error of the eye.
  Arms: Automated Refraction; Manual Refraction
Device: Phoropter — Manual refraction and ETDRS chart
  Arms: Refraction with a Hand-held Device Supported by Mobile App.
Device: Autorefractor — Automated refraction
  Arms: Refraction with a Hand-held Device Supported by Mobile App.

SUMMARY:
Single-center, open-label, prospective study in healthy volunteers desiring refraction for correction of visual acuity to compare a handheld device supported by a mobile application with the phoropter and autorefractor.

DETAILED DESCRIPTION:
Single-center, open-label, prospective study in healthy volunteers desiring refraction for correction of visual acuity to compare a handheld device supported by a mobile application with the phoropter and autorefractor in male or female subjects 30 to 65 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age 30 through 65 years at the time of consent
* Binocular vision
* Subject desires refraction for correction of visual acuity and vision can be corrected in each eye to 20/20 (LogMAR 0.0)
* Willing and able to give informed consent and follow all study procedures and requirements
* Ability to speak and understand the English language

Exclusion Criteria:

* Spherical correction > +8 or < -10
* Using anticholinergic medications (including first-generation antihistamines) or other medications known to affect visual acuity within the greater of 3 days or 5 half-lives prior to enrolling in this study
* Using an investigational drug or approved therapy for investigational use within the greater of 3 days or 5 half-lives prior to enrolling in this study
* Has initiated any new medication in the past 2 weeks that, in the best medical judgment of the investigator, would impact their participation in the study or ability to use the device
* Eye disease, including but not limited to:

  * Glaucoma (≥ 22 mmHg intraocular pressure)
  * Cataracts (≥ 1+ nuclear sclerotic cataract, ≥ 1+ cortical, posterior subcapsular cataract [any grade using the Lens Opacities Classification System III])
  * Macular degeneration (retinal pigmented epithelium mottling and/or any drusen within 500 μm of macula)
  * Eye infection (corneal ulcer, corneal infiltrates, superficial punctate keratitis)
  * Keratoconus
  * Diabetic neuropathy/retinopathy (≥ mild nonproliferative diabetic retinopathy)
  * Cytomegalovirus retinitis
  * Color blindness (any color deficiency)
  * Diabetic macular edema (evidence of fluid)
  * Amblyopia
  * Chronic or acute uveitis (cells and/or flare in anterior chamber)
  * Strabismus (exotropia, esotropia, and hypertropia)
  * Abnormal astigmatism (mild to severe, > 5 diopters)
  * Macular hole
* Eye surgery within the last 12 months (including Lasik or lens replacement)
* Subject does not have the physical dexterity to properly operate the device or the on the smartphone in the investigator's opinion.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Peace, MD, Principal Investigator — United Medical Research Institute
Locations (1):
- United Medical Research Institute, Inglewood, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: BCVA with handheld device with app.
  Phoropter: Manual refraction and ETDRS chart
  Autorefractor: Automated refraction
Period: Overall Study
Arm/Group | All Participants
Started | 230
Completed | 143
Not Completed | 87

BASELINE CHARACTERISTICS:
Arm/Group | Refraction With a Hand-held Device Supported by Mobile App.
Number analyzed (Participants) | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 230
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 115
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: BVCA Utilizing Refraction Results From Handheld Device Compared to Manual Refraction Methods for the Age Stratum 45 Through 65 Years
Description: Best-corrected visual acuity (BVCA) utilizing refraction results using the handheld device with supporting application will be compared to standard manual refraction methods (using a phoropter) for the age stratum 45 through 65 years.
Time Frame: Through study completion, an average of 5 months
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | All Participants
Number analyzed (Participants) | 143
logMAR
  BCVA handheld device | 0.06 [0.04 to 0.08]
  BCVA manual refraction | 0.02 [0 to 0.04]
  BCVA automated refraction | 0.03 [0.01 to 0.05]

ADVERSE EVENTS:
Time Frame: 6 months
Description: No difference from standard definition. None observed.
Arm/Group | Refraction With a Hand-held Device Supported by Mobile App.
All-Cause Mortality (participants affected / at risk) | 0/230
Serious Adverse Events (participants affected / at risk) | 0/230
Other Adverse Events (participants affected / at risk) | 0/230

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT03929588/Prot_SAP_000.pdf